CLINICAL TRIAL: NCT04231786
Title: Breast Ultrasonography Findings in Patients Over 30 Years With Polycystic Ovary Syndrome
Brief Title: Breast Ultrasonography and Polycystic Ovary Syndrome
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Pınar Kadirogulları, Pınar Kadiroğulları M.D, Department of Obstetrics and Gynecology,Principal Investigator, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: 2019.05.122
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Breast Diseases; Polycystic Ovary
Keywords: breast diseases; fibrocystic breast; polycystic ovari syndrome; fibroadenoma
MeSH Terms: conditions — Breast Diseases; Polycystic Ovary Syndrome; Cystic Fibrosis; Fibroadenoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Breast ultrasonography findings — Breast ultrasonography findings in patients over 30 years of age diagnosed with polycystic ovary syndrome.

SUMMARY:
The results of the evaluation of breast ultrasonography results of patients with polycystic ovary syndrome diagnosis over 30 years of age will be evaluated.

Patients admitted to the outpatient clinic and rotterdam criteria according to laboratory data and polycystic ovary syndrome patients diagnosed by the same radiologist the next day after the end of menstrual breast ultrasonography. The aim of this study is to show the association of polycystic ovary syndrome and fibrocystic breast.

ELIGIBILITY:
Inclusion Criteria:

* Over 30 years
* diagnosed with polycystic ovary syndrome according to rotterdam criteria
* no previous history of breast disease
* female patients

Exclusion Criteria:

* Under 30 years
* polycystic ovary syndrome
* patients with a previously known history of breast disease

Ages: 30 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: patients over 30 years of age diagnosed with polycystic ovary syndrome breast ultrasonography findings in these patients
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2020-07-14 (Actual); Study Completion 2020-07-14 (Actual)

PRIMARY OUTCOMES:
Breast ultrasonography findings | 1 month
  Breast ultrasonography findings in patients over 30 years of age diagnosed with polycystic ovary syndrome. THE PRESENCE OF FIBROCISTIC DISEASE WILL BE EVALUATED FOR FIBROADENOMA OR OTHER BREAST DISEASE. YES OR NO ; WILL BE REGISTERED.

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni Sultan Süleyman Training and Research Hospital, Istanbul, Turkey (Türkiye)